CLINICAL TRIAL: NCT00267059
Title: Lenalidomide (Revlimid) in Patients With Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Lenalidomide (Revlimid) in Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0175
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Chronic Lymphocytic Leukemia; Lenalidomide; Revlimid; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 10 mg/day, orally once a day for 28 days
  Other Names: CC-5013; Revlimid

SUMMARY:
The goal of this clinical research study is to learn if lenalidomide (Revlimid®) can help to control CLL in patients who have already received standard therapy. The safety of lenalidomide will also be studied.

DETAILED DESCRIPTION:
Lenalidomide is designed to change the body's immune system and may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete medical history and physical exam. Blood (between 2-4 teaspoons) and urine will be collected for routine tests. For patients taking Coumadin, blood will be collected (2-4 teaspoons) to measure anticoagulation in order to closely monitor your clotting ability for the purpose of adjusting your Coumadin dose, if necessary. This blood test is called an INR (International Standard Method to follow anticoagulation). You will have a bone marrow biopsy and aspirate. To collect a bone marrow biopsy and aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. These two collections are performed as one single procedure. You also will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart). Women who are able to have children must have a negative urine pregnancy test.

If you are found to be eligible to take part in this study, you will take lenalidomide by mouth every morning at about the same time for 28 days. This is considered 1 cycle. The dose and schedule of lenalidomide may be adjusted up or down depending on how your disease responds and the side effects you experience.

During this study, you will have blood samples (about 1 tablespoon each) taken once a week during the Cycle 1 until a stable dose of lenalidomide has been found. You will then have about 1 tablespoon of blood drawn every 2 weeks for an additional cycle and then once a month from then on while you are on study. Blood tests (about 1 tablespoon each) may be done more frequently if the dose of medication needs to be adjusted or if you experience side effects. Every month during the first 3 months, you will have a physical exam to see how you are doing. You will have a physical exam every 3 months from then on. After the first 3 months of treatment, a bone marrow biopsy and aspirate is going to be collected to evaluate your response to the treatment. In participants who continue to receive treatment, a bone marrow biopsy and aspiration are going to be repeated every 6 months during the first year, and then once a year after that while on study.

You will be required to return to M. D. Anderson at least once a month, for the first 3 months, and until a stable dose of lenalidomide has been established. Following this, you will be required to return at least every 3 months while taking the medication . Women who are able to have children must have a negative pregnancy test 10-14 days before the start of therapy and a repeat pregnancy test 24 hours before the start of lenalidomide, every week for the first 4 weeks, every 4 weeks if they have regular menstruation, every 2 weeks if their periods are irregular, and 30 days after they stop taking lenalidomide. Only if you have had a hysterectomy or no menstrual periods for at least 24 months in a row, will you not be required to have these pregnancy tests and use birth control.

You may continue to receive treatment as long as your disease is responding and no intolerable side effects occur. You will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for multiple myeloma. Lenalidomide use in chronic lymphocytic leukemia is considered experimental. Up to 45 patients may take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with B-cell CLL with indications for treatment by National Cancer Institute (NCI) Working Group Criteria, or Rai Stage III or IV or patients with CLL requiring treatment because of any of the following: disease related symptoms, progressive marrow failure (development or worsening of anemia and/or patients' thrombocytopenia) progressive splenomegaly, progressive lymphoadenopathy, progressive lymphocytosis
2. Patients who have received a minimum of one prior purine analog-based chemotherapy regimen. Prior treatment with corticosteroids, immunotherapy, monoclonal antibody or radiation therapy is permitted. All previous cancer therapy, including radiation, hormonal therapy and surgery must have been discontinued 2 weeks prior to treatment in this study. Any cytotoxic chemotherapy must be discontinued 4 weeks prior to treatment in this study.
3. Age more or equal to 18 years (CLL is not observed in patients less than 18 years of age).
4. Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status 0-2.
5. Adequate renal function indicated by serum creatinine less or equal to 2 and adequate hepatic function indicated as total bilirubin less or equal to 2 times the upper limit of normal.
6. Understand and sign Informed Consent after the investigational nature, study design, risks and benefits of the study have been explained.
7. Females of childbearing potential (FCBP)must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
8. Continued from #7. Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
9. Continued from #8. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
10. Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation can be enrolled in the study as long as they have a reasonable expectation to have been cured with treatment modality received.

Exclusion Criteria:

1. Known sensitivity to thalidomide or its derivatives
2. The development of erythema nodosum as characterized by a desquamating rash while taking thalidomide or similar drugs.
3. Prior use of lenalidomide
4. Concurrent use of other chemotherapy agents.
5. Known positivity for Human immunodeficiency virus (HIV) or infectious hepatitis type A, B or C.
6. Pregnant or lactating females.
7. A serious medical condition, laboratory abnormality or psychiatric illness that would pose the subject at unacceptable risk if he/she were to participate in the study or that would interfere with the ability of the patient to carry out the treatment program or confine the ability to interpret the data from the study.
8. Documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood).
9. Active cardiovascular disease as defined by the New York Heart Association class 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — UT M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Takahashi K, Hu B, Wang F, Yan Y, Kim E, Vitale C, Patel KP, Strati P, Gumbs C, Little L, Tippen S, Song X, Zhang J, Jain N, Thompson P, Garcia-Manero G, Kantarjian H, Estrov Z, Do KA, Keating M, Burger JA, Wierda WG, Futreal PA, Ferrajoli A. Clinical implications of cancer gene mutations in patients with chronic lymphocytic leukemia treated with lenalidomide. Blood. 2018 Apr 19;131(16):1820-1832. doi: 10.1182/blood-2017-11-817296. Epub 2018 Jan 22. PMID 29358183
- [Derived] Ferrajoli A, Lee BN, Schlette EJ, O'Brien SM, Gao H, Wen S, Wierda WG, Estrov Z, Faderl S, Cohen EN, Li C, Reuben JM, Keating MJ. Lenalidomide induces complete and partial remissions in patients with relapsed and refractory chronic lymphocytic leukemia. Blood. 2008 Jun 1;111(11):5291-7. doi: 10.1182/blood-2007-12-130120. Epub 2008 Mar 11. PMID 18334676
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 12/7/05 - 8/7/09; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Forty five patients were registered on this study. Forty four were evaluable. One patient never received treatment.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 19
Age Continuous [Median (Full Range); unit: years] | 63 [49 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Overall Response Categories
Description: Overall Response defined as participant had either complete response (CR) or partial response (PR) assessed after three cycles, at six months and yearly thereafter using the NCI-Working Group Criteria: Complete Response, Complete Response with Nodules, Partial Response, or No Response.
Time Frame: Evaluated after three 28-day cycles of lenalidomide.
Population: Analysis was intention to treat (ITT): Forty four patients received treatment.
Measure: Number; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 44
Participants
  Complete Response | 3
  Complete Response With Nodules | 1
  Partial Response | 10
  No Response | 30

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 24/44
Other Adverse Events (participants affected / at risk) | 34/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=44)
Pseudomonas Aeruginosa Bactremia (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pain (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Death (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9)
Pneumocystis carinii pneumonia (Infections and infestations) | 2 (2)
Mucormycosis (Gastrointestinal disorders) | 1 (1)
Fever of unknown origin (Infections and infestations) | 6 (6)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Rotavirus (Gastrointestinal disorders) | 1 (1)
Tumor Flare (General disorders) | 1 (1)
Secondary Malignancy Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)
Viral Hepatitis Reactivation (Immune system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Criptosporididosis (Gastrointestinal disorders) | 1 (1)
Prostate Infection (Infections and infestations) | 1 (1)
Stroke (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=44)
Neutropenia (Blood and lymphatic system disorders) | 13 (170)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (103)
Anemia (Blood and lymphatic system disorders) | 5 (72)
Fatigue (General disorders) | 14 (75)
Diarrhea (Gastrointestinal disorders) | 6 (50)
Rash (Skin and subcutaneous tissue disorders) | 12 (43)
Tumor Flare (General disorders) | 15 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No